# STUDY PROTOCOL

Version 1.0 – Date: September 9, 2025

| <b>Document Type:</b> Study Protocol | |
|---|---|
| <b>Official Title:</b> A Cross-Sectional Observational Study to Eval Depression, and Health-Related Quality of Life and Their Der in Adults With Type 2 Diabetes Attending an Outpatient Meta | nographic and Clinical Correlates |
| Sponsor: National Taiwan University Hospital | |
| <b>Principal Investigator:</b> Prof. Ching-Yuan Wang, MD, PhD, Department of Metabolism, National Taiwan University Hospital | |
| <b>Study Coordinator:</b> Yi-Chieh Chung, MSN, RN, Department of Metabolism, National Taiwan University Hospital | |
| NCT Number: Pending assignment | |
| <b>Protocol Version and Date:</b> Version 1.0 – September 9, 2025 | |
| IRB Approval: National Taiwan University Hospital REC – Approval No. 202508155RIND | |
| Study Site: Outpatient Metabolism Clinic, National Taiwan University Hospital, Taipei, Taiwan | |
| <b>Confidentiality Statement:</b> This document contains confidential information that must not be disclosed to anyone other than the study sponsor, investigators, and authorized regulatory authorities without prior written permission. | |
| Signatures | |
| Principal Investigator: | Date: |
| Study Coordinator: | Date: |

### 1. Study Summary

This study investigates the psychological well-being, depression severity, and health-related quality of life among adults with Type 2 Diabetes. It aims to identify demographic and clinical correlates that may influence these outcomes to inform integrated physical and psychological care strategies in diabetes management.

### 2. Study Design

This is a cross-sectional observational study conducted at a single site (National Taiwan University Hospital). Participants will complete standardized questionnaires during one outpatient visit. There is no follow-up period, and no intervention is administered.

### 3. Study Population

Eligible participants include adults (≥20 years old) diagnosed with Type 2 Diabetes attending the outpatient metabolism clinic. Exclusion criteria include inability to consent or complete questionnaires due to cognitive impairment or language barriers.

## 4. Sample Size

A total of approximately 500 participants are anticipated, based on feasibility and sufficient statistical power to detect medium effect sizes in multivariate analyses ( $\alpha = 0.05$ , power = 0.8).

#### 5. Data Collection Instruments

Participants will complete the following validated instruments:

- EQ-5D-5L for health-related quality of life.
- PHQ-9 for depression severity.
- Shalom Scale for psychological well-being.

In addition, demographic and clinical data (e.g., age, sex, education, diabetes duration, HbA1c, BMI, and complications) will be collected from medical records or self-report.

#### 6. Variables and Measures

Independent variables include demographic (age, sex, education, marital status, employment), and clinical variables (HbA1c, BMI, disease duration, complications).

Dependent variables include Shalom Scale total score (psychological well-being), PHQ-9 total score (depression severity), and EQ-5D-5L index and VAS (health-related quality of life).

### 7. Statistical Analysis Plan

Data will be analyzed using descriptive statistics, correlation analysis (Pearson's r), group comparisons (t-test or ANOVA), and multiple linear regression to identify predictors of psychological well-being.

All analyses will be performed using SPSS or R statistical software, with a significance level of 0.05.

### 8. Confidentiality and Data Protection

Participant information will be coded and de-identified. Only authorized research staff will have access to the key linking identifiers to data. Data will be stored securely in password-protected systems approved by the institution and retained for at least three years following study completion.

#### 9. Ethical Considerations

This study was reviewed and approved by the National Taiwan University Hospital Research Ethics Committee (Approval No. 202508155RIND). Participation is voluntary, and all participants will provide written informed consent. The study poses minimal risk as it involves only questionnaire completion and data collection from existing medical records.

#### 10. Contact Information

Principal Investigator: Prof. Ching-Yuan Wang, MD, PhD

Study Coordinator: Yi-Chieh Chung, MSN, RN

Department of Metabolism, National Taiwan University Hospital

Tel: +886-2-2312-3456

Email: yi-chieh.chung@ntuh.gov.tw

This English version is prepared for public posting on ClinicalTrials.gov under 42 CFR Part 11.